CLINICAL TRIAL: NCT04206943
Title: Phase I/ II Study of Cluster of Differentiation 19 (CD19) Specific CAR-T Cells (ISIKOK 19) in Relapsed/Refractory Acute Lymphoblastic Leukemia (ALL) and Non Hodgkin Lymphoma (NHL)
Brief Title: Study of CD19 Specific Chimeric Antigen Receptor Positive T Cells (CAR-T) in ALL and NHL
Acronym: ISIKOK-19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Collaborators: Acıbadem Atunizade Hospital (Other); The Scientific and Technological Research Council of Turkey (Other); Acıbadem Labcell (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD19-SP-CAR-T
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-09

CONDITIONS: Acute Lymphoblastic Leukemia; Non Hodgkin Lymphoma
Keywords: CAR-T Cell; CD19; ALL; NHL; Cancer; Chimeric Antigen Receptor
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Neoplasms | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Low Dose (Experimental): 4 x 10^6 Car-T cell/ kg
  Interventions: Biological: Car-T Cell Therapy
- B High Dose (Experimental): 6 x 10^6 Car-T cell/ kg
  Interventions: Biological: Car-T Cell Therapy

INTERVENTIONS:
Biological: Car-T Cell Therapy — Lymphodepletion Protocol:
  * -6. Day: Cyclophosphamide 300 mg / m^2 i.v.
  * -5. -4. and -3. Days: Fludarabine 30 mg / m^2 i.v. In addition, one day before the lymphodepletion protocol, xanthine oxidase enzyme inhibitor tablets received 100 mg / day p.o. and 0.9% sodium chloride solution 2000 ml / day i.v. infusion on protocol day received and continues for 2 weeks
  Car-T cells are administered in 3 split doses. Day 0: 20% or 40% (20% in patients with high tumor burden - in patients with bulky disease and / or more than 15% blast in bone marrow, 40% in patients with low tumor burden) Day 2: 30% or 50%, (the total amount of Car-T cell dose that should be given in the first 2 days should be 70%.) Third dose (%30);is given on the 7th day in the absence of cytokine release syndrome, or if cytokine release syndrome occurs, Car-T cells are given within 1 month if the number of copies falls below 5,000 / ml in 2 consecutive measurements.

SUMMARY:
It is a treatment that activates and strengthens the immune system against cancer. Recently, T cell receptors have been genetically rearranged by adaptive T cell therapies, which are promising in the fight against cancer, and are now able to recognize antigens on tumor cells. These modified T cell receptors are called chimeric antigen receptors. Many previous clinical studies have shown that different CAR-T cells are effective in relapse / refractory B cell cancers and NHL.

DETAILED DESCRIPTION:
Clinical trials of CAR-T cell therapy started at the end of 1990s. Phase I and II trials have still evaluated the efficacy and safety of CAR-T cells in hematological and solid cancers. The therapy involves drawing blood from patients and isolation of the T cells. Next, the T cells are genetically engineered in a laboratory by using virus or sleeping beauty to produce receptors on their surface named as chimeric antigen receptors. As the last step, the CAR-T cells are infused back into the patient. After infusion, it is expected that the CAR-T cells further increase in number in the patient's body and with the help of their engineered receptor to recognize and target the antigen on the surface of the cancerous cells for antitumor effect.

ELIGIBILITY:
Inclusion Criteria:

* Been diagnosed with CD19 (+) B-Acute lymphoblastic lymphoma or CD19 (+) Non-Hodgkin Lymphoma
* Having a measurable disease
* Relapsed/ refractory (at least 2 cases to the ward; in relapse after autologous transplantation in NHL) disease
* CD19 (+) expression in tumor cells by bone marrow/tissue or peripheral blood flow cytometry for relapse patients in the 3-month before the study period
* Bone marrow relapse after allogenic stem cell transplantation and at least 6 months between CAR-T (ISIKOK-19 ©) cell infusion and stem cell transplantation
* Philadelphia gene + B-ALL patient should have received second line treatment with tyrosine kinase inhibitor (TKI) or the usage of tyrosine kinase inhibitor (TKI) for the patient is contraindicated
* Patient; lack of appropriate donor, complications due to previous stem cell transplantation, or rejection of stem cell transplantation as a treatment option after consultation with a physician, or lack of allogenic stem cell transplantation due to high tumor burden.
* Lack of organ dysfunction:

  1. Maximum serum creatinine value: 1.7 mg / decilitre (male patients), 1.4 mg / decilitre (female patients)
  2. Liver function tests are within normal limits
  3. Bilirubin <2.0 mg / decilitre
  4. Central oxygen pressure in room air > 91% and no dyspnea
  5. Measurement of left ventricular ejection fraction ≥45% and left ventricular systolic function ≥28% by echocardiography during screening
* Expected survival is ≥ 3 months
* Performance condition: Karnofsky ≥ 50%
* Consent to oral contraceptives
* Approve treatment

Exclusion Criteria:

* Concomitant history of cardiac, hepatic, neurologic, nephrologic, psychiatric, autoimmune and additional oncological diseases affecting physiological functions
* Life expectancy <2 months
* Hepatitis B, Hepatitis C, Human immunodeficiency virus infection
* Before CAR-T (ISIKOK-19 ©) cell infusion

  1. Systemic steroid treatments, tyrosine kinase inhibitors, hydroxyurea, short-acting cytotoxic drugs should be stopped 72 hours before.
  2. 1 week ago, vincristine, 6-mercaptopurine, 6-thioguanine, methotrexate (if <25 mg / m^2), cytosine arabinoside (if <100 mg / m^2), asparaginase and intrathecal treatments should be stopped.
  3. 2 weeks ago, salvage treatments (chemotherapy drugs other than lymphodepletion as part of the protocol, clofarabine, cytosine arabinoside (if> 100 mg / m^2), anthracyclines, methotrexate (if ≥25 mg / m^2), drugs used for graft versus host disease, long-acting growth factors, vincristine, immunomodulatory drugs should be stopped.
  4. Radiotherapy taken outside the central nervous system should be stopped 2 weeks prior.
  5. Any systemic treatment with pegylated asparaginase and donor lymphocyte infusion should be stopped 4 weeks prior.
  6. Anti-t cell therapies containing T cell lysis or toxic antibodies should be stopped 8 weeks before.
  7. Radiotherapy for the central nervous system should be stopped 8 weeks ago.
  8. Less than 3 months after stem cell transplantation
  9. Below 60% in tissue biopsies and / or CD19 expression in tumor cells by flow cytometric analysis in bone marrow is below 85%
* Allergic to drugs that are used at any stage of treatment
* Having received experimental drug treatment in the last month
* Previously entered a cellular therapy and / or a gene therapy program
* Disapproval of the storage of tissues and cells
* Isolated disease that occurs outside the bone
* A genetic disease associated with concomitant bone marrow failure
* Active Grade 2-4 acute or diffuse chronic graft versus host disease
* Being pregnant or breastfeeding
* Disapproval the treatment
* Patients with slow CAR-T cell expansion (the cell number is not doubled in 48 hours) and with less than 10% expression of CAR-T cells during production, < 60% cytotoxicity results in in-vitro study (i.e, patients whose product is inappropriate)

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-10-12 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 6 Months
  Type, frequency and severity of adverse events (AEs) and laboratory abnormalities.

SECONDARY OUTCOMES:
Complete Remission Rate | 3 Months
  It is determined by the evaluation of complete remission (CR) obtained in the first 3 months.
Total Response Rate | 3 Months
  CR obtained in the first 3 months is determined by evaluation of partial remission, incomplete partial remission and stable disease responses.
Duration of Remission (DOR) | 6 Months
  Duration of remission (DOR) is defined as the duration from the date when the response criteria of CR or CRi is first met to the date of relapse or death due to underlying cancer, whichever occurs first.
Relapse Free Survival (RFS) | 6 Months
  Relapse free survival (RFS) is measured by the time from achievement of CR or CRi whatever occurs first to relapse or death due to any cause during CR or CRi.
Progression Free Survival | 6 Months
  Only in the NHL is the duration from CAR T cell infusion to progression
Event-Free Survival (EFS) | 6 Months
  Event free survival (EFS) is the time from date of first Car-T cell infusion to the earliest of the following:
  * Death from any cause
  * Relapse
Overall Survival | 6 Months
  Overall survival (OS) is the time from date of first Car-T Cell infusion to the date of death due to any reason.
Duration to maximum response | 6 Months
  The duration from date of the first Car-T cell infusion to complete remission in ALL.
  The duration from date of the first Car-T cell infusion to complete remission and partial remission in NHL
The impact of baseline tumor burden on response | 6 Months
  Best overall response will be summarized by baseline tumor burden (MRD, extramedullary disease, etc.)
The relationship between CRS/CRES efficiency | 6 Months
  The relationship between CRS / CRES grades and total response rates are determined by correlation between DOR, RFS, EFS, PFS, OS.
The relationship between the total response and Car-T Cell persistence | 6 Months
  The relationship between total response and the number of Car-T copies is determined by the correlation between DOR, RFS, EFS, PFS, OS
The relationship between Car-T Cell product content and responses | 6 Months
  The relationship between Car-T Cell subgroups and total response are determined by the correlation between DOR, RFS, EFS, PFS, OS.
Car-T cell proliferation capability | 6 months
  The relationship between the Car-T Cell proliferation capability and the total response, are determined by the correlation between DOR, RFS, EFS, PFS, OS.
The relationship between MRD grade and clinical response | 6 Months
  The relationship between MRD grade and total response are determined by correlation between DOR, RFS, EFS, PFS, OS.
The relationship between the incidence of immune response to Car-T cells and the persistence of Car-T cell | 6 Months
  It is assessed as the relationship between antiserum effectivity against Car-T cells and Car-T cell copy number in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Ercument Ovali, MD, Study Director — Director
Locations (1):
- Acıbadem Labcell Cellular Therapy Laboratories, Istanbul, Turkey (Türkiye)